CLINICAL TRIAL: NCT03130738
Title: Dose-Ranging Study of the Efficacy and Safety of Miconazole Oil Used for 7 or 14 Days Compared With Vehicle in the Treatment of Otomycosis
Brief Title: Dose-Ranging Study for Miconazole Oil for Treatment of Otomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hill Dermaceuticals, Inc. (Industry)
Collaborators: QST Consultations, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD-MCZ-PHII-DRF062016
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Results first posted 2020-05-08 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis | interventions — Miconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, investigators, and study staff will not be masked as to the treatment duration assigned to each subject (7 versus 14 days). For subjects receiving the 14-day treatment with study drug, the contents of the study drug (active versus placebo) will be masked to the subject, investigator, and study staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 7-Day Miconazole Oil (Miconazole 2%) (Active Comparator): 7 days of 2x per day of treatment with Miconazole Oil (Active Drug Product 2% Miconazole)
  Interventions: Drug: 7-Day Miconazole Oil (Miconazole 2%)
- 14-Day Miconazole Oil (Miconazole 2%) (Active Comparator): 14 days of 2x per day of treatment with Miconazole Oil (Active Drug Product 2% Miconazole)
  Interventions: Drug: 14-Day Miconazole Oil (Miconazole 2%)
- 14-Day Placebo - Oil Vehicle (Placebo Comparator): 14 days of 2x per day of treatment with Placebo - Oil Vehicle, Study Drug base without active ingredient
  Interventions: Drug: 14-Day Placebo - Oil Vehicle

INTERVENTIONS:
Drug: 7-Day Miconazole Oil (Miconazole 2%) — 7 days of 2x per day treatment with Miconazole Oil (Active Drug Product 2% Miconazole)
  Other Names: Miconazole
  Arms: 7-Day Miconazole Oil (Miconazole 2%)
Drug: 14-Day Miconazole Oil (Miconazole 2%) — 14 days of 2x per day treatment with Miconazole Oil (Active Drug Product 2% Miconazole)
  Other Names: Miconazole
  Arms: 14-Day Miconazole Oil (Miconazole 2%)
Drug: 14-Day Placebo - Oil Vehicle — 14 days of 2x per day treatment with Placebo - Oil Vehicle, Study Drug base without active ingredient
  Other Names: (Miconazole) Placebo Oil Vehicle
  Arms: 14-Day Placebo - Oil Vehicle

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of active treatment (miconazole oil) for 7 versus 14 days, and to compare 14 days of active treatment (miconazole oil) to inactive treatment (placebo) over a 14-day treatment duration, in subjects with fungal infection (otomycosis) of the external ear.

DETAILED DESCRIPTION:
Miconazole, an imidazole antifungal agent, is commonly used for different types of fungal skin infections, such as Candida, ringworm, jock itch, athlete's foot, nail fungus, vaginal yeast infections, and oropharyngeal candidiasis. The 2% formulation of miconazole is commonly used for dermatophytic infections. The mechanisms of action of miconazole against fungi in general appear to be applicable to fungi associated with otomycosis, in that miconazole has been demonstrated to have activity in vitro against some clinical isolates of fungi associated with human otomycosis in the US.

Miconazole targets the cytochrome P450-dependent enzyme 14-α-sterol demethylase, an enzyme that is also involved in mammalian cholesterol synthesis, resulting in inhibition of ergosterol biosynthesis in the cell membrane of the fungal organism. Because ergosterol is an important component of the cell membrane, inhibition of its synthesis inhibits fungal cell growth.

In addition to its activity toward the enzyme 14-α-sterol demethylase, miconazole also leads to increased reactive oxygen species in fungal organisms, which appears to result in fungicidal activity.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated otomycosis of the external ear only, age more than 2 year

Exclusion Criteria:

* Pregnancy
* Other dermatoses or conditions of the ear that may interfere with the evaluation of otomycosis, including concomitant otic infections (including bacterial infection) that require antimicrobial treatment, disease that has spread beyond the external ear(s), or pre-existing skin atrophy of the affected ear(s)
* Tympanostomy tube or perforated tympanic membrane in the ear(s) that will be treated
* Previous surgery affecting the ear(s) that will be treated, except for prior tympanostomy tube(s) that had been removed and had completely healed
* Previous use of medicated treatments for otomycosis or participation in another investigational study within 28 days of study entry
* Previous use of any systemic antifungal therapy, warfarin, and immunosuppressive or immune-stimulating drugs within 28 days of study entry, or systemic steroids within 3 months of study entry
* Recurrent otomycosis that had been unresponsive to previous antifungal treatment
* Known hypersensitivity to any of the components in the test formulation

Min Age: 25 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosario G Ramirez, MD, Study Director — Hill Dermaceuticals, Inc.; Jack Wazen, MD, Principal Investigator — Silverstein Institute; Quyen T Nguyen, MD, Principal Investigator — UCSD; Kenneth Hodge, MD, Principal Investigator — Advanced ENT and Allergy; Kenneth S Maxwell, MD, Principal Investigator — Piedmont Ear, Nose and Throat Associates; Woo Linda, MD, Principal Investigator — Head and Neck Surgery Specialists
Locations (6):
- United States (6):
  - Head and Neck Surgery Specialist, Chula Vista, California
  - University of California San Diego, La Jolla, California
  - Ear Nose and Throat Associates of Southe Florida, Boynton Beach, Florida
  - Silverstein Institute, Sarasota, Florida
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Piedmont ENT Associates, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 7-Day Miconazole Oil (Miconazole 2%) | 14-Day Miconazole Oil (Miconazole 2%) | 14-Day Placebo - Oil Vehicle
Started | 23 | 22 | 20
Completed | 20 | 20 | 14
Not Completed | 3 | 2 | 6

BASELINE CHARACTERISTICS:
Population: Baseline participants from ITT population which consisted of subjects entered and randomized, by randomized group. ITT population includes MITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | 7-Day Miconazole Oil (Miconazole 2%) | 14-Day Miconazole Oil (Miconazole 2%) | 14-Day Placebo - Oil Vehicle | Total
Number analyzed (Participants) | 23 | 22 | 20 | 65
Age, Continuous [Median (Full Range); unit: years] | 64.0 [11 to 84] | 66.0 [8 to 86] | 62.5 [20 to 85] | 64 [11 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 32
  Male | 13 | 11 | 9 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 22 | 20 | 18 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 21 | 18 | 16 | 55
  More than one race | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 22 | 20 | 65
Mycological culture [Count of Participants; unit: Participants]
  Positive mycological culture | 12 | 12 | 14 | 38
  Negative mycological culture | 11 | 10 | 6 | 27
Pruritus - investigator assessed [Count of Participants; unit: Participants]
  Mild, moderate or severe | 10 | 11 | 14 | 35
  None | 13 | 11 | 6 | 30
Debris [Count of Participants; unit: Participants]
  Scant, moderate or Heavy | 12 | 12 | 14 | 38
  None | 11 | 10 | 6 | 27
Presence of fungal elements [Count of Participants; unit: Participants]
  Present | 12 | 12 | 14 | 38
  Absent | 11 | 10 | 6 | 27
Pain [Count of Participants; unit: Participants]
  Present | 9 | 10 | 11 | 30
  Absent | 14 | 12 | 9 | 35

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint
Description: Percentage of subjects in MITT population, at the "Test of Cure" visit with "Therapeutic cure", defined as a negative fungal culture plus "clinical cure" defined as the absence of all otomycosis signs and symptoms for pruritus, debris, fungal elements, and pain.
Time Frame: At Test of Cure visit (Day 15 for 7 Day Active and Day 22 for 14 Day Active and 14 Day Vehicle)
Population: Actual number of participants analyzed under Primary efficacy endpoint are MITT population, defined as subjects who had a clinical diagnosis of otomycosis confirmed by positive fungal culture.
Measure: Count of Participants; unit: Participants
Arm/Group | 7-Day Miconazole Oil (Miconazole 2%) | 14-Day Miconazole Oil (Miconazole 2%) | 14-Day Placebo - Oil Vehicle
Number analyzed (Participants) | 12 | 12 | 14
Participants | 1 | 3 | 1

2. Secondary Outcome: Secondary Efficacy Endpoints
Description: 1. Percentage of subjects in MITT population with clinical cure at the Test of Cure Visit
  2. Percentage of subjects in MITT population with a negative fungal culture at the Test of Cure Visit
  3. Percentage of subjects in MITT population with a negative fungal culture at the Test of Cure visit as well as individual sign or symptom score of 0 or 1 on each of the scales for pruritus and debris and a score of 0 on each of the scales for fungal elements and pain (Secondary therapeutic cure).
  4. Percentage of subjects in MITT population with individual signs or symptoms with a score of 0 or 1 on each of the scales for pruritus and debris and a score of 0 on each of the scales for fungal elements and pain (Secondary clinical cure).
Time Frame: At Test of Cure visit (Day 15 for 7 Day Active and Day 22 for 14 Day Active and 14 Day Vehicle)
Population: Percentage of subjects in the MITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | 7-Day Miconazole Oil (Miconazole 2%) | 14-Day Miconazole Oil (Miconazole 2%) | 14-Day Placebo - Oil Vehicle
Number analyzed (Participants) | 12 | 12 | 14
Participants
  Clinical Cure | 2 | 4 | 2
  Negative Fungal Culture | 4 | 5 | 3
  Secondary Therapeutic Cure | 3 | 5 | 1
  Secondary Clinical Cure | 7 | 6 | 4

ADVERSE EVENTS:
Time Frame: The study duration for each subject was up to 30 days (up to 14 days of treatment, and 8 days of follow-up, including the visit window of up to 8 additional days after the scheduled day to complete the final visit), starting from entry and randomization in the study. Start at Screening Visit and ends at final visit which is the Test of cure visit.
Description: AEs were recorded and classified using MedDRA terminology. All treatment-emergent adverse events (TEAEs), defined as any AE with onset on or after date of first study drug application, summarized by drug group, number of subjects reporting TEAE, system organ class, preferred term, severity, relationship to study drug, and seriousness. Each subject counted once within a system organ class or preferred term using event with the highest severity and greatest relationship within each classification.
Arm/Group | 7-Day Miconazole Oil (Miconazole 2%) | 14-Day Miconazole Oil (Miconazole 2%) | 14-Day Placebo - Oil Vehicle
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 9/23 | 10/22 | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7-Day Miconazole Oil (Miconazole 2%) (N=23) | 14-Day Miconazole Oil (Miconazole 2%) (N=22) | 14-Day Placebo - Oil Vehicle (N=20)
Ear pain. Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (4)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
discharge. discomfort. erosion. pain. pruritus. site pain (General disorders) | 4 (4) | 6 (8) | 9 (12) — administration site conditions
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
site infection. ear fugal infection. myringitis.bacterial otitis externa. otitis media. skin infecti (Infections and infestations) | 4 (4) | 3 (4) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
arthritis. rheumatoid arthritis. (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proprietary Information will need prior written consent of the sponsor. PI will hold in confidence and not disclose any Proprietary Information unless disclosure has its prior written consent from sponsor, or that the information is disclosed to personnel who need to know. Sponsor will not prohibit PI to comply with applicable laws and regulations, provided PI gives prior written notice to Sponsor. Disclosure allowed if legally required and accorded confidential treatment.

DOCUMENTS (2):
  • Study Protocol (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT03130738/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT03130738/SAP_001.pdf